CLINICAL TRIAL: NCT06971237
Title: Response Assessment for Advanced HCC of Combined SIRT and Immunotherapy Treatment
Brief Title: SIRT and Peri-immunotherapy : a New Concept
Acronym: IMSIRT
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241625; IDRCB (Other: 2024-A02309-38)
Record Dates: First submitted 2025-04-25; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC), Classified as BCLC Stage B or C, Treated With a Combination of Selective Internal Radiation Therapy
Keywords: Hepatocellular Carcinoma; Advanced Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Atezolizumab ± Bevacizumab and Yttrium-90 Radioembolization — Atezolizumab ± Bevacizumab: Peri-immunotherapy with , with or without bevacizumab, given before and after SIRT.
  - Yttrium-90 Radioembolization: Selective Internal Radiation Therapy (SIRT) via intra-arterial injection of Yttrium-90 microspheres for liver tumor control
Drug: Atezolizumab ± Bevacizumab — Standard systemic immunotherapy administered without SIRT, using atezolizumab with or without bevacizumab.

SUMMARY:
The combination of selective internal radiation therapy (SIRT) with immunotherapy represents an innovative and potentially highly effective therapeutic strategy for the treatment of advanced-stage hepatocellular carcinoma (BCLC stage B or C). Although promising results have been observed in preliminary clinical trials, further research is needed to better understand the underlying mechanisms, optimize treatment protocols, and confirm the long-term efficacy and safety of this combined approach

DETAILED DESCRIPTION:
This retrospective cohort study aims to evaluate the efficacy and safety of a novel combination treatment for advanced hepatocellular carcinoma (HCC), involving Selective Internal Radiation Therapy (SIRT) with Yttrium-90 (Y90) microspheres and peri-immunotherapy (atezolizumab ± bevacizumab) administered in both neoadjuvant and adjuvant settings. The study targets patients with Barcelona Clinic Liver Cancer (BCLC) stage B or C HCC, initially deemed ineligible for curative therapies such as resection, transplantation, or percutaneous ablation.

Recent advances in immunotherapy have shown promise for HCC treatment, but overall response rates remain low due to the immunosuppressive tumor microenvironment. SIRT delivers high-dose localized radiation directly to the tumor, inducing immunogenic cell death and potentially priming the immune system for enhanced response to immune checkpoint inhibitors. This study investigates whether this combination can produce synergistic anti-tumor effects, prolong progression-free survival (PFS) and overall survival (OS), and potentially downstage tumors to make curative treatment feasible.

Data will be retrospectively collected from electronic health records (Orbis), imaging systems (PACS), and pathology databases at the AP-HP GH Paris-Saclay institutions (Hôpital Paul Brousse and Hôpital Bicêtre). A total of 60 patients treated between 2021 and 2024 will be included. Key clinical variables (e.g., age, sex, comorbidities, AFP), imaging response (based on RECIST 1.1, mRECIST, iRECIST, LI-RADS criteria), treatment parameters (e.g., Y90 dose, immunotherapy schedule), histological findings, and adverse events (CTCAE grading) will be systematically extracted and anonymized.

A matched control group of patients treated with immunotherapy alone will be used for comparative analysis. Imaging will be reviewed independently by two senior abdominal imaging radiologists. Statistical analyses will be conducted using R Software (version 3.2.3) in collaboration with the GH Paris-Saclay methodology unit.

This study complies with French and European data protection regulations (MR-004) and has obtained ethical approval from the Bicêtre ethics committee (CER POLETHIS). Patients are informed by mail and included upon non-objection within one month.

The overarching goal is to determine whether the SIRT + peri-immunotherapy protocol offers improved disease control and survival outcomes compared to standard treatment, while maintaining acceptable safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Diagnosis of hepatocellular carcinoma (HCC) confirmed by imaging or biopsy Tumor > 6 cm Child-Pugh score A to B7 Not eligible for curative treatment (resection, ablation, transplant, TACE) Macrovascular invasion or AFP > 100 ng/mL Treated with intra-arterial Yttrium-90 SIRT combined with atezolizumab ± bevacizumab

Exclusion Criteria:

Age < 18 Non-HCC diagnosis on imaging or pathology Child-Pugh > B7 Prior immunotherapy or intra-arterial hepatic treatment Under legal guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced hepatocellular carcinoma (BCLC stage B or C), not eligible for curative treatments, treated with SIRT and/or immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Tumor Response Rate | At 3, 6, 9 and 12 months post-treatment
  Proportion of patients achieving complete or partial response, evaluated by CT or MRI using RECIST 1.1, mRECIST, iRECIST, and LI-RADS therapeutic criteria

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From treatment to disease progression or death, up to 12 months
  Time between start of treatment and first documented progression or death, based on imaging and clinical records
Overall Survival (OS) | From treatment to death, up to 12 months
  Time from treatment initiation to death from any cause.
Treatment-Related Adverse Events | through study completion, an average of 1 year
  Assessment of adverse events related to SIRT and/or immunotherapy, graded using CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Maïté Lewin, Professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Paul Brousse
Locations (1):
- Hôpital Paul Brousse - Radiology Department, Villejuif, France

IPD SHARING:
Plan to Share IPD: No